CLINICAL TRIAL: NCT04251572
Title: Hepatitis C Reinfection After Successful Directly Acting Antiviral Treatment: A Belgian Interventional Multicenter Study
Brief Title: HCV Reinfection After DAA Therapy in PWID in Belgium
Acronym: REINF_HCV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other); Jessa Hospital (Other); Algemeen Ziekenhuis Vesalius (Other); CAD Limburg (Unknown); Sint-Trudo (Unknown); Free Clinic Antwerp (Unknown); Ziekenhuis Netwerk Antwerpen (ZNA) (Other); Clinique Saint Joseph, Liège (Other); Centre Hospitalier Universitaire Saint Pierre (Other); Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Principal Investigator, Geert Robaeys, Principal Investigator, Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18/0012U
Record Dates: First submitted 2018-05-30; First posted 2020-02-05 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Hepatitis C Virus Infection, Response to Therapy of; Drug Use
MeSH Terms: conditions — Hepatitis C | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HCV reinfection after DAA therapy in PWID (Experimental): Hepatitis C virus reinfection after directly acting antiviral treatment in persons who inject drugs. DAA therapy is an inclusion criteria, not an intervention.
  Interventions: Other: Blood sampling; Other: questionaires

INTERVENTIONS:
Other: Blood sampling — Blood sampling
Other: questionaires — Included participants will complete a baseline questionnaire at end of treatment (EOT) and a follow-up questionnaire throughout the follow-up period (Table 1). The questionnaires collect information on socio-demographics (age, gender, ethnicity, employment status, education level, housing status, incarceration, medical history and OST), injecting drug use (drugs injected, injection frequency and sharing of needle/syringe, cookers, cotton/filter or water). Details on the received DAA regime including mode of administration (direct observed therapy, pill box, etc.) and self-reported data on treatment adherence will also be recorded.

SUMMARY:
The primary aim of this study is to calculate the incidence of HCV reinfection after successful DAA treatment among people who have recently injected drugs. The secondary aim is to identify factors associated with reinfection in this population.

Individuals with active injecting drug abuse with a chronic HCV infection who have achieved end of treatment response (ETR; defined as non-detectable HCV RNA at end of treatment) to any interferon-free DAA combination will be included in this multicenter interventional study.

DETAILED DESCRIPTION:
This protocol is an adapted version of the protocol 'Hepatitis C reinfection after successful directly acting antiviral treatment: A North-Atlantic multicenter interventional study'. The investigators will plan this study so that the data are similar to this protocol and results can be compared within this alliance of hepatologists with special interest in care for substance users.

Study schedule: Data collection will be performed according to the study schedule shown in Table 1. Following assessment for SVR12, participants will be followed for 2 years at 6 months' intervals at the discretion of each study site.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age 18 years or older
* Injecting drug use within 6 months before start of treatment
* Achieved an ETR following at least eight weeks of DAA treatment
* Completed DAA treatment no more than 6 months prior to inclusion
* Blood sample drawn within 6 months pre-treatment stored at -70° C

Exclusion Criteria:

* Patients not fulfilling the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of reinfections in people who inject drugs after cure for hepatitis C infection with direct antiviral therapy | up to two years
  Number of reinfections with hepatitis C per 100 persons

SECONDARY OUTCOMES:
questionnaire to Identify risk factors associated with HCV reinfection | day 1
questionaire to Identify risk factors associated with HCV reinfection | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Geert Robaeys, prof. dr., Principal Investigator — Hasselt University; Rob Bielen, dr., Study Chair — Hasselt University
Locations (10):
- Belgium (10):
  - Free Clinic Antwerp, Antwerp
  - ZNA Stuivenberg, Antwerp
  - CHU Saint-Pierre, Brussels
  - Ziekenhuis Oost-Limburg, Genk
  - AZ Maria-Middelares, Ghent
  - CAD Limburg, Hasselt
  - Jessa Ziekenhuis, Hasselt
  - CHC Saint-Josephe, Liège, Liège
  - Sint-Trudo Ziekenhuis, Sint-Truiden
  - AZ Vesalius, Tongeren

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Busschots D, Bielen R, Koc OM, Heyens L, Verrando R, de Galocsy C, Van Steenkiste C, Nevens F, Midgard H, Dalgard O, Robaeys G. Hepatitis C reinfection in former and active injecting drug users in Belgium. Harm Reduct J. 2021 Oct 12;18(1):102. doi: 10.1186/s12954-021-00552-x. PMID 34641896